CLINICAL TRIAL: NCT02360553
Title: The Effect of Internet Based Intervention (OBESEGO!) Towards Obesity Among Adolescents
Brief Title: The Effect of ObeseGO! Towards Adolescent Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: azmawati
Record Dates: First submitted 2015-02-05; First posted 2015-02-10 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Adolescent Behavioral Change

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): ObeseGO!-web-based intervention
  Interventions: Behavioral: ObeseGO!
- Control (Other): Given pamphlets education mainly on diet and physical activity
  Interventions: Behavioral: Pamphlets material

INTERVENTIONS:
Behavioral: ObeseGO! — The intervention group were received the obeseGO! intervention which is an internet-based intervention. The participants and the parents who are randomly chosen to enroll in this intervention group were provided with the ObeseGO! website. The website was accessed at www.obesego.com. The website consists of various informations on healthy lifestyle, diet and ways to overcome obesity.
  Arms: Intervention
Behavioral: Pamphlets material — The control group will be given pamphlets material on diet and physical activity.
  Arms: Control

SUMMARY:
Adolescents nowadays is having most of their times other than school hours spending on screen by playing games, watching the movies and surfing the internet. Thus, it was suggested that Internet-based interventions have the potential for establishing healthy dietary style and physical activity that may persist in adulthood and reduce the risk of chronic disease. Preventing adolescent obesity requires an attitude of willingness by adolescents to implement healthy behaviors. By providing the health related activities in website, it would help the adolescents to spend time on screen by having something which can benefit them and improve their knowledge and attitudes.

DETAILED DESCRIPTION:
This study done in improving the health promotion in Malaysia. It will be an evidenced in creating the most effective way in creating the awareness among adolescent. By having an effective health promotion it will help in reducing the prevalence of obesity and improving health among adolescents hence will reducing the comorbidities among adulthood.

ELIGIBILITY:
Inclusion Criteria:

* Students aged of 16 years old (adolescents) in secondary school in Kuala Lumpur who have BMI of more than 25 kg/m2, have one guardian or parent who willing to join the study and having access to internet at home were then selected to join this study

Exclusion Criteria:

* those who are having existing medical condition and having weight loss more than 2 kg in last two months

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Body mass index | 3 months
  reduce of BMI

SECONDARY OUTCOMES:
Waist Circumference | 3 months
Body fat percentage | 3 months